CLINICAL TRIAL: NCT05901714
Title: An Open-label, Single-sequence, Drug-drug Interaction Study in Healthy Participants to Assess the Effect of Phenytoin on the Pharmacokinetics of a Single Oral Dose of Afimetoran (BMS-986256) (Part 1) and the Effect of Steady-state Afimetoran on the Pharmacokinetics of Midazolam (Part 2)
Brief Title: A Study to Assess the Effect of Phenytoin on the Drug Levels of Afimetoran and the Effect of Afimetoran on the Drug Levels of Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IM026-026
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Healthy Participants
Keywords: BMS-986256; Afimetoran; Midazolam; CYP3A4; Phenytoin
MeSH Terms: interventions — Phenytoin; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Afimetoran followed by phenytoin + afimetoran (Experimental)
  Interventions: Drug: Afimetoran; Drug: Phenytoin
- Part 2: Midazolam followed by afimetoran + midazolam (Experimental)
  Interventions: Drug: Afimetoran; Drug: Midazolam

INTERVENTIONS:
Drug: Afimetoran — Specified dose on specified days
  Other Names: BMS-986256
Drug: Phenytoin — Specified dose on specified days
  Arms: Part 1: Afimetoran followed by phenytoin + afimetoran
Drug: Midazolam — Specified dose on specified days
  Arms: Part 2: Midazolam followed by afimetoran + midazolam

SUMMARY:
This study will consist of 2 parts. The study will evaluate whether administration of phenytoin impacts the single-dose drug levels of afimetoran and BMT-271199 (Part 1) and will evaluate whether multiple administrations of afimetoran impact the drug levels of midazolam and 1-hydroxymidazolam (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 19.0 kilograms per meter squared (kg/m^2) to 32.0 kg/m2, inclusive, and body weight ≥ 55 kg, at screening.

Exclusion Criteria:

* Any significant acute or chronic medical illness or any other condition listed as a contraindication in the phenytoin (Part 1) or midazolam (Part 2) package inserts.
* History of seizure (including simple febrile seizure), epilepsy, severe head injury (including concussion), multiple sclerosis, or other known neurological condition which the investigator considers to be clinically significant.
* Current or recent (within 3 months of study intervention administration) GI disease that could impact upon the absorption of study intervention.

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 53 days
  Parts 1 and 2
Area under the plasma concentration-time curve from time zero to time of the last quantifiable concentration (AUC[0-T]) | Up to 53 days
  Parts 1 and 2
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC[INF]) | Up to 53 days
  Parts 1 and 2

SECONDARY OUTCOMES:
Time to attain maximum observed plasma concentration (Tmax) | Up to 53 days
  Parts 1 and 2
Terminal half-life (T-Half) | Up to 53 days
  Parts 1 and 2
Apparent total body clearance of the drug from the plasma (CLT/F) | Up to 53 days
  Parts 1 and 2
Number of participants with adverse events (AEs) | Up to 124 days
  Parts 1 and 2
Number of participants with clinical laboratory abnormalities | Up to 66 days
  Parts 1 and 2
Number of participants with physical examination abnormalities | Up to 66 days
  Parts 1 and 2
Number of participants with vital sign abnormalities | Up to 66 days
  Parts 1 and 2
Number of participants with electrocardiogram (ECG) abnormalities | Up to 66 days
  Parts 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT05901714.html